CLINICAL TRIAL: NCT05687734
Title: Outcome of Reconstruction of Failed and Neglected Terrible Triad Injury of the Elbow
Brief Title: Outcome of Failed and Neglected Terrible Triad Injury of the Elbow
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mo'men Moustafa Mohamed Saber, Doctor, Assiut University
Other Study IDs: Outcome of elbow injury
Record Dates: First submitted 2022-12-15; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Elbow Injury
MeSH Terms: conditions — Elbow Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate the results of reconstruction of neglected and failed cases of terrible triad of the elbow

DETAILED DESCRIPTION:
A terrible triad injury consists of posterior dislocation of the elbow associated with a radial head fracture and a coronoid fracture. This injury occurs during a fall onto an outstretched arm, and it presents a disruption of the bony and capsuloligamentous structures from the lateral side, which progresses anteriorly and medially.The primary goal of surgical treatment for terrible triad injury is to restore elbow function with. good stability. The current standard treatment involves internal fixation and reconstruction of the bony and ligamentous structures to allow early mobilization. Fixation or replacement of radial head fractures and lateral ligament reconstruction represent the main operative procedures. A biomechanical and clinical study showed that restoration of the coronoid process and anterior capsule is an important step for a stable elbow. old "terrible triad" of elbow with no operative history is difficult to treat. The elbow's functions and stabilization can be recovered by thorough elbow release, repair of coronoid process and anterior capsule, radial head fixation or replacment reconstruction or repaire of, lateral collateral ligament and reinsertion of the common extensor tendon, combined with hinged external fixator Although improved knowledge of this injury has yielded favourable clinical outcomes, complications continue to occur, including stiffness, recurrent subluxation or dislocation, heterotopic ossification, ulnar nerve neuropathy, and arthritis.The common causes of revision after terrible triad injury reconstruction are stiffness and recurrent instability, Stiffness and instability, among all these complications, are indeed the most recurring. A stiff or unstable elbow is very poorly tolerated because of the lack of compensatory motion in adjacent joints, So it's very important to detect causes and risk factors that leading to fail terrible triad reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* • Age from 15 to 70 years' old

  * Neglected cases more than 4 weeks
  * Early failed cases whom had any intervention whether conservative treatment as cast or hinged elbow brace etc or operative and still complaining of instability of the elbow. In less than 6 weeks
  * Late Failed cases whom had any intervention whether conservative treatment as cast or hinged elbow brace etc or operative and still complaining of instability of the elbow after more than 6 weeks .

Exclusion Criteria:

* • Older than 70 years old and younger than 15 years old

  * Nerve injury
  * Associated soft tissue loss
  * Patients needs Total Elbow Replacement or Arthrodesis

Ages: 15 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: • All cases fulfilling the Inclusion and Exclusion Criteria admitted to Assuit university over two year from the beginning of the study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The final end results will be assessed according to degree of improvement according to DASH score performance index | DASH score assessment preoperative and at 4,8 weeks 6 months and 1 year postoperative.Follow up:2 weeks postoperative for stitches removal, 6 weeks by x ray to assess reunion, 3 and 6 months by x ray to assess reunion.1 year by MSCT to assess reunion
  The final end results will be assessed according to degree of improvement according to DASH score performance index (The disability of the arm, shoulder and hand)(is an upper-extremity specific outcome measure that was introduced by the American Academy of Orthopedic Surgeons in collaboration with a number of other organizations)(The main part of the DASH is a 30-item disability/symptom scale concerning the patient's health status during the preceding week. The items ask about the degree of difficulty in performing different physical activities because of the arm, shoulder, or hand problem (21 items), the severity of each of the symptoms of pain, activity-related pain, tingling, weakness and stiffness (5 items), as well as the problem's impact on social activities, work, sleep, and self-image (4 items). Each item has five response options. The scores for all items are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability).

CONTACTS AND LOCATIONS:
Overall Officials: Aly Mohamden Mohamed, Professor, Study Director — Assiut University; Waleed Riad Saleh, Professor, Study Director — Assiut University

REFERENCES:
- [Background] Kachooei AR, Mellema JJ, Tarabochia MA, Chen N, van Dijk CN, Ring D. Involvement of the lesser sigmoid notch in elbow fracture dislocations. J Shoulder Elbow Surg. 2016 Oct;25(10):1571-6. doi: 10.1016/j.jse.2016.02.013. Epub 2016 May 24. PMID 27233485
- [Background] Giannicola G, Calella P, Piccioli A, Scacchi M, Gumina S. Terrible triad of the elbow: is it still a troublesome injury? Injury. 2015 Dec;46 Suppl 8:S68-76. doi: 10.1016/S0020-1383(15)30058-9. PMID 26747922
- [Background] Zhang J, Tan M, Kwek EBK. Outcomes of coronoid-first repair in terrible triad injuries of the elbow. Arch Orthop Trauma Surg. 2017 Sep;137(9):1239-1245. doi: 10.1007/s00402-017-2733-8. Epub 2017 Jun 20. PMID 28634742
- [Background] Fitzgibbons PG, Louie D, Dyer GS, Blazar P, Earp B. Functional outcomes after fixation of "terrible triad" elbow fracture dislocations. Orthopedics. 2014 Apr;37(4):e373-6. doi: 10.3928/01477447-20140401-59. PMID 24762843
- [Background] Ritali A, Rotini R, Cavallo M, Marinelli A, Guerra E. Instability/stiffness in elbow fracture dislocation. Lo Scalpello-Journal. 2020 Mar 22;34:30-5.
- [Background] Sun Z, Li J, Luo G, Wang F, Hu Y, Fan C. What constitutes a clinically important change in Mayo Elbow Performance Index and range of movement after open elbow arthrolysis? Bone Joint J. 2021 Feb;103-B(2):366-372. doi: 10.1302/0301-620X.103B2.BJJ-2020-0259.R3. PMID 33517717